CLINICAL TRIAL: NCT05919277
Title: A Dengue Sero-prevalence Study in the Metropolitan Area of Buenos Aires
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Fundacion GESICA (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: DENGUE SEROPREVALENCE IN AMBA
Record Dates: First submitted 2023-06-13; First posted 2023-06-26 (Actual); Last update posted 2023-09-13 (Actual); Status verified 2023-09

CONDITIONS: Dengue; Flavivirus Infections
MeSH Terms: conditions — Dengue; Flavivirus Infections

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Dengue Immunoglobulin G antibodies performed with ELISA — All participants who agree to participate by signing an informed consent form will undergo a finger prick for the determination of Immunoglobulin G antibodies measured by ELISA. In a subgroup of persons who test positive, they will be invited to have blood drawn for neutralization determination in order to study serotypes and the presence of other flaviviruses.

SUMMARY:
The objective of this observational study of dengue seroprevalence in the metropolitan area of Buenos Aires is to know what percentage of the population has antibodies against dengue in persons 18 years of age or older who are residents of the city of Buenos Aires or its metropolitan area. The main questions to be answered are:

* What is the seroprevalence of antibodies against dengue measured by Immunoglobulin G determination by ELISA
* Characterize the different dengue serotypes in the affected population. Participants will undergo a small blood draw to determine the presence of Immunoglobulin G antibodies against dengue.
* Tests will also be performed to determine infection by flaviviruses other than dengue virus.

DETAILED DESCRIPTION:
A two-stage stratified design will be used. The primary sampling units will be mostly defined as the census sections of the 2010 National Census of Population, Households and Dwellings. It has 5 strata, constructed through a functional relationship between the income quintiles obtained in the Annual Household Survey (AHS) and the variables that were surveyed in the census. Stratum 1 corresponds to the lowest income population, while stratum 5 corresponds to the highest. The first stage of sampling in this framework will consist of about 100 to 300 primary sampling units, called primary units areas, selected with a probability proportional to size, the measure of size being the total number of dwellings.

A sample of 1,487 dwellings is proposed. In each primary unit area, a number of dwellings will be selected to be visited by enumerators, who will make a list of all members residing in the dwelling (regardless of whether they are from the same household) and select a member aged ≥18 years to proceed with the survey. This last selection is a 3rd and final sampling stage that will define the sample of 1487 participants to be tested. The sample size was calculated based on the estimated probability of pre-infection for each of the municipalities and localities participating in the survey.

ELIGIBILITY:
Inclusion Criteria:

* - Age ≥18 at the time of signing the informed consent.
* - Resident of the Buenos Aires metropolitan area

Exclusion Criteria:

* To be ≤17 years old.
* Inability to give informed consent.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: A two-stage stratified design will be used. The primary sampling units will be mostly defined as the census tracts of the 2010 national population, household and housing census. It has 5 strata, constructed through a functional relationship between the income quintiles obtained in the Annual Household Survey (HHS) and variables that were surveyed in the census. Stratum 1 is the lowest income population, while stratum 5 corresponds to the highest. The first stage of sampling in this framework will be made up of nearly 100 to 300 primary sampling units, called UP areas, selected with probability proportional to size, the measure of size being the total number of dwellings. A sample size of 1487 dwellings is proposed.
Sampling Method: Probability Sample
Enrollment: 1487 (Estimated)
Dates: Start 2023-09-11 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2024-09 (Estimated)

PRIMARY OUTCOMES:
Seroprevalence | Through study completion, an average of 1 year
  Percentage of the population with Immunoglobulin G antibodies against dengue fever

SECONDARY OUTCOMES:
Other flavivirus prevalence | Through study completion, an average of 1 year
  Percentage of population with Immunoglobulin G antibodies to dengue, but found to be cross-reactive to other flaviviruses on plaque neutralization.
Specific dengue serotype | Through study completion, an average of 1 year
  Dengue-specific serotype among the Immunoglobulin G-positive population.

CONTACTS AND LOCATIONS:
Overall Officials: Alejandro Macchia, MD, Study Director — Fundacion GESICA
Locations (1):
- Fundación GESICA, Ciudad Autónoma de Buenos Aire, Buenos Aires, Argentina

IPD SHARING:
Plan to Share IPD: No